CLINICAL TRIAL: NCT04717050
Title: Reducing Metabolic Dysregulation in Obese Latina Breast Cancer Survivors Using Physical Activity: The ROSA Trial
Brief Title: Reducing Metabolic Dysregulation in Obese Latina Breast Cancer Survivors Using Physical Activity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-221
Record Dates: First submitted 2021-01-19; First posted 2021-01-20 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Coronary Artery Disease; Stroke; Type2 Diabetes
Keywords: Breast Cancer; Coronary Artery Disease; Stroke; Type2 Diabetes; Exercise Therapy
MeSH Terms: conditions — Breast Neoplasms; Coronary Artery Disease; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive combine training (PCT) (Experimental): Participants will be randomly assigned to Progressive combine training (PCT) group.
  Participants will have two (2) baseline tests, then begin a two phase PCT program.
  * Phase 1: Supervised 16-week resistance and cardiovascular exercise at a local YMCA (months 1-4) or remotely at home via Zoom
  * Participants will receive midpoint testing, approximately week 8.
  * Phase 2: Unsupervised 16-week resistance and cardiovascular exercise at a local YMCA (months 5-8) or remotely at home
  * Participants will receive midpoint testing, approximately two months into phase 2.
  After the two (2) 16-week phases, participants will be followed for 4 months.
  Interventions: Behavioral: Progressive combine training (PCT)
- Attention Control (AC) (Active Comparator): Participants will be randomly assigned to Attention Control (AC) group.
  Two (2) baseline tests will be performed prior to starting the program. Participants will perform 12 months of home-based stretching and have a 1x test performed during months 2, 4, 6, 8 and 10. Two (2) tests will be performed in month 12.
  Interventions: Behavioral: Attention Control (AC)

INTERVENTIONS:
Behavioral: Progressive combine training (PCT) — 8 month exercise program with 4 month follow up.
  Arms: Progressive combine training (PCT)
Behavioral: Attention Control (AC) — 12 month stretching program
  Arms: Attention Control (AC)

SUMMARY:
This study is about testing whether exercise will improve fitness and lessen risk factors related to heart disease, diabetes, and obesity in Latina breast cancer survivors.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied. The purpose of this research is to determine whether a 16-week exercise program will improve fitness and lessen risk factors related to coronary artery disease, stroke, and type 2 diabetes in patients who have breast cancer and is sustainable for a Latina population to incorporate into their lifestyle following completion of the 16-week intervention.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

Participants in this study will be randomly assigned into one of the study groups: Progressive Combine Training (PCT) or Attention Control.

* Progressive combined training (PCT) will be performed in 2 phases:

  1. supervised 16-week resistance and cardiovascular exercise at a local YMCA (months 1-4) or remotely at home via Zoom.
  2. unsupervised 16-week resistance and cardiovascular exercise at a local YMCA (months 5-8) or remotely at home with weekly check-ins with trainer.
* Attention Control Group: 51 weeks home-based stretching

All participants will undergo seven blood draws and participate in nine testing visits.

Participation is expected to last 12 months for all participants.

It is expected that about 160 people will take part in this research study.

The American Cancer Society is supporting this research study by providing funding for the research study.

ELIGIBILITY:
Inclusion Criteria:

* Women newly diagnosed (Stage I-III) breast cancer.
* Over the age of 18 years; children under the age of 18 will be excluded due to rarity of disease
* The effects of exercise on the developing fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.
* Are centrally obese with the following criteria[84] (determined by study team at eligibility screening): BMI >30 kg/m2 (calculated using height and weight; an upper limit BMI will not be set; we will rely on obtaining physicians' clearance to assess full eligibility) or body fat >30% (estimated by bioelectrical impedance), and waist circumference >35 in.
* Have undergone a lumpectomy or mastectomy.
* Have received and completed neoadjuvant or adjuvant chemotherapy and/or radiation therapy within the past 12 months.
* Speak English or Spanish
* Self-identify as Latina
* Is in breast cancer remission with no detectable disease present
* Able to initiate a supervised exercise program (free from any cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity)
* Free from history of chronic disease including uncontrolled diabetes, hypertension or thyroid disease
* Have not experienced a weight reduction ≥10% within the past 6 months
* Currently participate in less than 60 minutes of structured exercise/week
* No planned reconstructive surgery with flap repair during trial and follow-up period
* May use adjuvant endocrine therapy if use will be continued for duration of study intervention
* Does not smoke (no smoking during previous 12 months)
* Willing to travel to Dana-Farber Cancer Institute for necessary data collection
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection, uncontrolled diabetes, hypertension or thyroid disease; women using Metformin to manage diabetes will be excluded from the trial
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* Patients with other active malignancies are ineligible for this study.
* Patients with metastatic disease
* Is not centrally obese as defined above
* Has not completed surgery, chemotherapy, or radiation treatment associated with their diagnosis
* History of any musculoskeletal, cardiorespiratory or neurological diseases that preclude the participation in exercise
* Participates in more than 60 minutes of structured exercise/week
* Is planning reconstructive surgery with flap repair during trial and follow-up period
* Currently smokes
* Is unable to travel to Dana-Farber Cancer Institute and/or exercise facility for necessary data collection
* Weight reduction ≥ 10% within past 6 months
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in Metabolic Dysregulation (MetD) After Completion of Phase 1 Progressive Combine Training (PCT) -Insulin Resistance | 16 weeks
  Changes from baseline in insulin resistance (IR) measured by Homeostasis Model Assessment (HOMA)
Change in Metabolic Dysregulation (MetD) After Completion of Phase 1 Progressive Combine Training (PCT) -Visceral adiposity | 16 weeks
  Changes from baseline in visceral adiposity (VA) measured by dual-energy X-ray absorptiometry (DXA), waist to hip ratio (WHR) and bioelectrical impedance technology (BIA)
Change in Metabolic Dysregulation (MetD) After Completion of Phase 1 Progressive Combine Training (PCT) -metabolic syndrome (MSY) | 16 weeks
  Frequency of metabolic syndrome (MSY) diagnosed by criteria accepted by the American Heart Association (AHA)

SECONDARY OUTCOMES:
Compare Metabolic Dysregulation (MetD) in Progressive Combine Training (PCT) and Attention (AC) groups -Insulin Resistance | 16 weeks
  Compare changes from baseline in insulin resistance (IR) measured by Homeostasis Model Assessment (HOMA) in Progressive Combine Training (PCT) and Attention (AC) groups
Compare Metabolic Dysregulation (MetD) in Progressive Combine Training (PCT) and Attention (AC) groups - Visceral adiposity | 16 weeks
  Compare changes from baseline in Visceral adiposity (VA) measured by dual-energy X-ray absorptiometry (DXA), waist to hip ratio (WHR) and bioelectrical impedance technology (BIA) in Progressive Combine Training (PCT) and Attention (AC) groups
Compare Metabolic Dysregulation (MetD) in Progressive Combine Training (PCT) and Attention (AC) groups - metabolic syndrome (MSY) | 16 weeks
  Compare frequency of metabolic syndrome (MSY) diagnosed by criteria accepted by the American Heart Association (AHA) in Progressive Combine Training (PCT) and Attention (AC) groups - metabolic syndrome (MSY)
Metabolic Dysregulation (MetD) Status During 4 month follow up period - insulin resistance (IR) | 16 weeks
  Change in insulin resistance (IR) status from end of study PCT to 4 month follow up measured by Homeostasis Model Assessment (HOMA).
Metabolic Dysregulation (MetD) Status During 4 month follow up period - Visceral adiposity (VA) | 16 weeks
  Change in Visceral adiposity (VA) status from end of study PCT to 4 month follow up measured by dual-energy X-ray absorptiometry (DXA), waist to hip ratio (WHR) and bioelectrical impedance technology (BIA).
Metabolic Dysregulation (MetD) Status During 4 month follow up period - metabolic syndrome (MSY) | 16 weeks
  Change in metabolic syndrome (MSY) frequency from end of study PCT to 4 month follow up diagnosed by criteria accepted by the American Heart Association (AHA)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu